CLINICAL TRIAL: NCT04347772
Title: Intensive Perioperative Nutrition Therapy
Brief Title: Effectiveness of Intensive Perioperative Nutrition Therapy Among Adults Undergoing Gastrointestinal & Oncology Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Zalina Abu Zaid, Principal Investigator, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 43546
Record Dates: First submitted 2019-11-20; First posted 2020-04-15 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-05

CONDITIONS: Perioperative Complication
Keywords: Perioperative Nutrition Therapy; Surgical Patients; Post-operative complication
MeSH Terms: interventions — Nutrition Therapy

STUDY DESIGN:
Intervention Model Description: This is a pragmatic randomized clinical trial involving patients undergoing major elective surgery.
  Baseline will be commenced before operation, when the decision to operate electively was made in the outpatient setting, and ended 6 hours before surgery. Next visit will be commenced on the first day that the patient was able to take free fluids or a light diet after operation, and ended 4 weeks after discharge from hospital.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplements Group - SS (Experimental): The SS will be received tailored and more intensive and ongoing nutrition support and lifestyle advice as compared with the NN and will be supplemented with ONS, available in 400g/can, providing 226 kcal/serving and 9.6 g protein/serving. Participants will be encouraged to consume the ONS in small, frequent, in between meals.
  All participants will receive standard post-operative care from clinical and nurse staff with commencement of free fluids and reintroduction of normal diet without interference by the researcher or protocol. The postoperative course will be carefully monitored. While complications will be noted as major or minor by using validated criteria (Buzby et al., 1988).
  Interventions: Dietary Supplement: Oral Nutrition Support
- Control Group - NN (No Intervention): While participants in NN which referred as control group will received the standard care of the clinic without supplemented with ONS. Nutritional advice will be based on a guideline specifically focused on treatment of symptoms such as nausea, vomiting, loss of appetite and diarrhoea, and how to deal with the symptoms through nutritional approaches. Basically, the advice will be given by the oncologist or nurses in the clinic.
  All participants will receive standard post-operative care from clinical and nurse staff with commencement of free fluids and reintroduction of normal diet without interference by the researcher or protocol. The postoperative course will be carefully monitored. While complications will be noted as major or minor by using validated criteria (Buzby et al., 1988).

INTERVENTIONS:
Dietary Supplement: Oral Nutrition Support — Intensive Nutrition Intervention
  Arms: Supplements Group - SS

SUMMARY:
Perioperative malnutrition is common in patients undergoing gastrointestinal and oncological surgery and it also associated with longer hospital stays, reduced responses to and increased complications from therapies, increased costs, poorer quality of life and lower survival rate. Evidence has shown that appropriate perioperative nutrition therapy have a significantly improve perioperative outcomes. Current practice emphasises the roles of early nutrition therapy as early intervention in order to combat the post-operative complications of patients and the implementation is now widely adopted. However, there is very limited data to date on the effects of perioperative nutrition therapy in patients before hospital admission, during hospital stay and after discharge to prevent the post-operative complications. Therefore, there is a need to study in this area in order to determine the effects of perioperative nutrition therapy to overcome the post-operative complications in patients undergoing surgery. This is a pragmatic randomized clinical trial will be conducted among sixty eight adults patient undergoing major elective surgery in Hospital Serdang. Participants will be randomized to one of two groups by means of sealed envelope into Intervention Group (SS) or Control Group (NN). All data will be collected during a face to face interview, blood sampling and direct anthropometric measurement with the participants at Hospital Serdang. The effects of intervention between treatment groups on outcome parameters will be carried out by using the SPSS General Linear Model (GLM) for repeated measure procedure. The perioperative nutrition therapy intervention implemented in the study will serve as a baseline data for providing an appropriate nutritional management in patients undergoing surgery.

DETAILED DESCRIPTION:
Malnutrition is well reported and common in surgery patients. Surgery itself leads to inflammation corresponding with the extent of the surgical trauma, and leads to a metabolic stress response. The existing research suggests that patients undergoing surgery for upper gastrointestinal or colorectal cancer are particularly at risk of malnutrition. Recent research from Malaysia shows almost similar findings from previous studies which is about 29.1% of surgical patients were malnourished and shows increase length of hospital stay, higher rate of surgical site infection and mortality.

Nutrition requirement for surgery is higher if compared with normal requirement in order to support speedy recovery. However, most of the patients especially cancer patients do unable to achieve even 50% energy requirement before operation. This will cause further depletion of nutritional status of patient. In conjunction with this, patients with suboptimal nutritional status pre-operatively will have a higher risk of postoperative complications. Interestingly, one of Malaysian study shows significant number of post-surgery complications compared to pre-surgery which was associated to the poor level of nutrition. The success of surgery does not depend exclusively on technical surgical skills but also on metabolic intervention therapy, taking into account the ability of patient to carry a metabolic load and to provide appropriate nutrition support. In fact, in patient with cancer, management during perioperative period may be crucial for long term outcome.

Nutrition therapy is the provision of nutrition or nutrients either orally (regular diet, therapeutic diet, e.g. fortified food, oral nutritional supplements) or via enteral nutrition (EN) or parenteral nutrition (PN) to prevent or treat malnutrition. Dietary advice or nutrition counselling is part of a nutrition therapy. In the surgical patient, the indications for nutritional therapy are prevention and treatment of catabolism and malnutrition. This affects mainly the perioperative maintenance of nutritional state in order to prevent postoperative complications. It is strongly recommended not to wait until severe disease-related malnutrition has developed, but to start nutrition therapy early, as soon as a nutritional risk becomes apparent.

Early oral feeding is the preferred mode of nutrition for surgical patients. Avoidance of any nutritional therapy bears the risk of underfeeding during the postoperative course after major surgery. Considering that malnutrition and underfeeding are risk factors for postoperative complications, early enteral feeding is especially relevant for any surgical patient at nutritional risk, especially for those undergoing upper gastrointestinal surgery e.g. for cancer. In addition, appropriate perioperative nutrition therapy has been shown on improvement of perioperative outcomes especially in gastrointestinal and oncologic surgical patients.

Early nutrition intervention or perioperative EN is optimising patient's nutritional status so that their bodies can receive optimal effects during surgical. The general indications for nutritional support therapy in patients undergoing surgery are the prevention and treatment of undernutrition, i.e. the correction of undernutrition before surgery and the maintenance of nutritional status after surgery, when periods of prolonged fasting and/or severe catabolism are expected. Morbidity, length of hospital stay, and mortality are considered principal outcome parameters when evaluating the benefits of nutritional support.

According to The European Society for Clinical Nutrition and Metabolism (ESPEN) Guidelines 2017, perioperative EN support will be indicated, when patient is unable to eat for more than 7 days preoperatively and in patient who cannot maintain oral intake more than 60-75% of recommended intake for more than 10 days. In addition, to most gastrointestinal surgeons, pre-operative nutritional support refers to a period of administration of supplementary calories, by enteral or parenteral route, prior to performing surgery in order to correct malnutrition and reduce the incidence of post-operative complications.

Maintenance or improvement in nutrition status is the key goal of medical nutrition therapy for individuals undergoing surgery. Although many patients tolerate therapy well and experience few or no post-operative complication, malnutrition is still a common condition, which affects quality of life and survival for many patients. To maintain or improve nutritional status, all barriers associated with oral intake should be aggressively addressed unless aggressive intervention is not warranted. Nutrition intervention are purposely-planned actions designed with the intent of changing behaviour, risk factor, environmental condition, or the aspect of health status for an individual, a target group, or the general population. The intervention involves dietetic strategies and strategies to meet the needs of surgical patients, which concentrate on helping patients to maintain and/or improve nutritional intake in the presence of symptoms, regain body weight or minimise weight loss and reduce post-operative complications.

Normally, the personalised dietetic intervention consists of strategies to modify the amount of food taken, either through advice or by provision of additional foods as snacks, fortification of foods to increase the energy and nutrient content; and the prescription of oral nutritional supplements. Ravasco and colleagues (2005) suggested that this type of intervention should be promptly carried out as early as possible as soon as any risk is identified and in close collaboration with the patient, along with monitoring of compliance to the diet.

Patients undergoing major surgery showed a consistently high prevalence of pre-operative malnutrition (50 -80%) and it is associated with higher post-operative mortality, morbidity, cost and longer hospital stay. Patients with severe nutritional risk in surgical patients with oral feeding, some improvements were shown in shortened duration of hospital stay and flatus, and some of wound and infectious complications. Particularly decreased hospital stay in patients is significant for prevention of increasing further complications and reduction in burden of hospital stay costs.

Studies show high prevalence of malnutrition or high nutritional risk during hospital admission but this is rarely assessed in the clinical setting especially patients who will undergone elective surgery. Surprisingly, a study in Latin American countries showed that nutrition information was included in the medical records of only 23% of patients and that 9% of patients received nutrition therapy, whereas up to 50% of patients were malnourished. Globally, hospital malnutrition is under-recognised, under-diagnosed and under-treated by health care professional, which may potentially of omission of nutritional assessments in routine patient assessment on admission. The use of nutrition screening tools i.e. Malnutrition Screening Tool (MST) or Nutritional Risk Screening (NRS) to identify surgical patient at risk of malnutrition are still low in Malaysian hospital setting. Currently, patient who has been scheduled to go for surgery will be admitted to the ward only two to three days prior to the operation date. Some of them are not screened and referred to dietitian for nutritional status assessment and intervene malnutrition before operation. Even these patients at risk of malnutrition or malnourished prior to the surgery. Two to three days admission prior to operation date is not enough to optimise their nutritional status when patient is having poor oral intake. And most of the time, surgery treatment needs to be delayed due to the nutritional status of these patients are not optimised prior surgery.

The use of oral nutritional supplementation (ONS), together with voluntary food intake, as a means of providing nutritional support to surgical patients is more straightforward; these products are easy to administer, comparatively cheap, free from complication and, with the range of flavours now available, palatable. Importantly, postoperative ONS has been shown to have a beneficial effect on outcome after surgery. Most studies have investigated the effect of nutrition therapy to look into the post-operative complication which ONS were prescribed during the pre-operative but not after the surgery. Conversely, there are limited data on the effects of perioperative nutrition therapy before and after surgery especially in Malaysia. Therefore, further research on the process of nutrition management, from screening/assessment on admission to nutritional support and monitoring needs to be conducted in this area in order to find good practices and should be mandated in routine patient care regardless of disease type.

ELIGIBILITY:
Inclusion Criteria:

* Those who receiving elective major surgery treatments
* Aged from 18 years old to 80 years old
* Malaysian
* Able to communicate verbally
* MST score ≥ 2
* Provided and signed informed consent

Exclusion Criteria:

* Those who had received pre-operative enteral or PN
* Those who requiring emergency surgery
* Complicated with chronic diseases and fluid retention (renal/ cardiovascular/ pulmonary/ hepatic)
* Those who participated in other research study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Length of Bowel function | 2 months
  To compare the effect of intensive perioperative nutrition therapy versus usual care on the length of bowel function. The duration of bowel start function post-operatively in hours or days will be recorded. The duration covers from zero hours after surgery until the first day of bowel function presented. The start of bowel function is the first day of commencement of any type of fluids or solid food given
Length of solid food toleration | 2 months
  To compare the effect of intensive perioperative nutrition therapy versus usual care on the length of solid food toleration. The duration of solid food toleration post-operatively in hours or days will be recorded. The duration covers from zero hours after surgery until the first day of reintroduction of solid food.
Length of hospital stay | 2 months
  To compare the effect of intensive perioperative nutrition therapy versus usual care on the length of hospital stay. The duration of hospital stay in days will be recorded. The duration covers from the day of ward admission (before operation) until discharge (after operation).

SECONDARY OUTCOMES:
Malnutrition Status - The scored Patient Generated Subjective Global Assessment (PG-SGA) | 2 months
  To examine malnutrition status in gastrointestinal and oncologic surgical patients in intervention group versus control group via Scored PG-SGA©. It consisted of two sections with seven domains. The first section, completed by the participant, is comprise of weight, food intake, symptoms, activities, as well as function. The second section will be completed by the researcher as it covered the disease and its relation to nutritional requirements, determination of metabolic demands, and followed by a nutrition-related physical examination. PG-SGA© scores that ranged from 0-35 reflected a greater risk of malnutrition. These scores will be transformed into global ratings - Stage A, B and C-which represented the states of being well-nourished, moderately malnourished, and severely malnourished, respectively. Data will be collected during baseline and at the end of visit.
Functional status - handgrip strength | 2 months
  To examine functional status in gastrointestinal and oncologic surgical patients in intervention group versus control group. Handgrip strength will be measured on the non-dominant hand using Jamar hand dynamometer. Subjects will be sat with their shoulder adducted and neutrally rotated, elbow flexed at 90º, forearm in neutral position, and standard verbal instructions will be given to the subjects to squeeze the dynamometer as hard as possible for three times after an interval of 5 seconds in between grips. Average of three successive attempts will be used as the final result.
Nutritional status - Body Mass Index (BMI) | 2 months
  To examine nutritional status in gastrointestinal and oncologic surgical patients in intervention group versus control group through BMI. Body weight and height will be taken with participants being shoeless and wearing lightweight clothing with empty pockets, without watches, or other accessories. Weight will be determined to the nearest 0.1 kg using a digital weighing scale. The machine will be calibrated every morning with a standard weight before it will be used. Height will be measured in the standing position to the nearest 0.1 cm using a SECA 206 microtoise tape which will be attached to the wall. All measurements will be taken twice by the same investigators, and the average will be used. Weight and height of the participants will be then used to calculate BMI. Data will be collected at baseline, first and at the end of visit.
Nutritional status - Mid Arm Circumference (MAC) | 2 months
  To examine nutritional status in gastrointestinal and oncologic surgical patients in intervention group versus control group through Mid Arm Circumference (MAC). MAC will be taken without any sleeve at measured arm, watches or other accessories. Subject is in a relaxed standing position with the arms hanging by the sides. MAC will be measured in the middle arm (same distant) from acromiole and radiale bone, to the nearest 0.1 cm using SECA 201 circumference measuring tape (SECA, British Indicators Ltd., United Kingdom). The caliper will be calibrated every morning before it will be used to minimize error during measurement. All anthropometric measurements will be taken twice by the same investigators, and the average will be used. Data will be collected at baseline, 1st and at the end of visit.
Nutritional status - Tricep Skinfold (TSF) | 2 months
  TSF will be taken without any sleeve at measured arm, watches or other accessories. Subject is in a relaxed standing position with the arms hanging by the sides. MAC will be measured first to determine the location of TSF measurement. TSF will be measured at the most posterior part of the triceps when viewed from the side at MAC level, to the nearest 0.1 mm using Harpenden skinfold caliper. The caliper will be calibrated every morning before it will be used to minimize error during measurement.All anthropometric measurements will be taken twice by the same investigators, and the average will be used. Data will be collected at baseline, 1st and at the end of visit.
Nutritional status - Serum Albumin | 2 months
  To examine nutritional status in gastrointestinal and oncologic surgical patients in intervention group versus control group by serum albumin. Data on serum albumin level will be obtained from patients' medical report at baseline and at the end of visit.
Nutritional status - Serum white blood cell | 2 months
  To examine nutritional status in gastrointestinal and oncologic surgical patients in intervention group versus control group by serum white blood cell (WBC). Data on WBC level will be obtained from patients' medical report at baseline and at the end of visit.
Nutritional status - Serum Haemoglobin | 2 months
  To examine nutritional status in gastrointestinal and oncologic surgical patients in intervention group versus control group by serum haemoglobin (Hb). Data on Hb level will be obtained from patients' medical report at baseline and at the end of visit.
Nutritional status - Serum C-reactive protein (CRP) | 2 months
  To examine nutritional status in gastrointestinal and oncologic surgical patients in intervention group versus control group by serum C-reactive protein (CRP). 10 ml of venous blood will be taken following overnight fast. The samples will be separated immediately by means of centrifugation (1800g for 10 min at 4°C). The serum will be stored at -80°C until analysis for the measurement of C-reactive protein which will be performed after all samples are collected. Serum C-reactive protein will be measured using the latex photometric immunoassay. Blood sample for CRP will be taken at baseline and at the end of visit.
Nutritional status - Dietary Intake | 2 months
  To examine nutritional status in gastrointestinal and oncologic surgical patients in intervention group versus control group by dietary intake. Dietary intake will be measured through a 24-hour dietary recall at baseline and two days of 24-hour dietary records during visit 1 & 3. Details of food information and descriptions, which included brand names, preparation and cooking methods, as well as recipes of any mixed dishes eaten during the study period, will be also recorded. Both groups will be provided an explanation by the researcher on how to record their 2-days intake in a food diary. They will be also given a detailed set of instructions together with a food album. The food album lists commonly consumed food and includes details of portion sizes to facilitate recalls of serving size and improve accuracy. A computerized local dietary analysis program, Nutritionist Pro version 2.0 will be used to analyze the nutrient intakes of the patients.

CONTACTS AND LOCATIONS:
Overall Officials: Zalina Abu Zaid, PhD, Principal Investigator — University Putra Malaysia
Locations (1):
- Hospital Serdang, Kajang, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: No
Sociodemographics data

REFERENCES:
- [Result] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Result] Smedley F, Bowling T, James M, Stokes E, Goodger C, O'Connor O, Oldale C, Jones P, Silk D. Randomized clinical trial of the effects of preoperative and postoperative oral nutritional supplements on clinical course and cost of care. Br J Surg. 2004 Aug;91(8):983-90. doi: 10.1002/bjs.4578. PMID 15286958
- [Result] MacFie J, Woodcock NP, Palmer MD, Walker A, Townsend S, Mitchell CJ. Oral dietary supplements in pre- and postoperative surgical patients: a prospective and randomized clinical trial. Nutrition. 2000 Sep;16(9):723-8. doi: 10.1016/s0899-9007(00)00377-4. PMID 10978851
- [Result] Kabata P, Jastrzebski T, Kakol M, Krol K, Bobowicz M, Kosowska A, Jaskiewicz J. Preoperative nutritional support in cancer patients with no clinical signs of malnutrition--prospective randomized controlled trial. Support Care Cancer. 2015 Feb;23(2):365-70. doi: 10.1007/s00520-014-2363-4. Epub 2014 Aug 6. PMID 25091056
- [Result] Jie B, Jiang ZM, Nolan MT, Zhu SN, Yu K, Kondrup J. Impact of preoperative nutritional support on clinical outcome in abdominal surgical patients at nutritional risk. Nutrition. 2012 Oct;28(10):1022-7. doi: 10.1016/j.nut.2012.01.017. Epub 2012 Jun 5. PMID 22673593
- [Derived] A'zim AZA, Zaid ZA, Yusof BNM, Jabar MF, Shahar ASM. Effectiveness of intensive perioperative nutrition therapy among adults undergoing gastrointestinal and oncological surgery in a public hospital: study protocol for a pragmatic randomized control trial. Trials. 2022 Nov 26;23(1):961. doi: 10.1186/s13063-022-06898-2. PMID 36435838